CLINICAL TRIAL: NCT04230655
Title: The Effects of a Low Energy Diet Versus Low Energy Diet and Intragastric Balloon in Adults With Obesity, All in Combination With Group Treatment: a Randomized, Controlled Trial
Brief Title: Weight Loss in Adults With Obesity Using a Combination of Low Energy Diet, Group Treatment and Intragastric Balloon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 256841
Record Dates: First submitted 2019-12-30; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Weight Loss; Non-Alcoholic Fatty Liver Disease
Keywords: Obesity; Weight loss; Low energy diet; Intragastric balloon; Group treatment; Non-alcoholic fatty liver disease; Quality of life; Body weight; Glucose metabolism; Eating behavior; Microbiomics; Physical activity; Gastrointestinal symptoms; Psychological parameters
MeSH Terms: conditions — Obesity; Weight Loss; Non-alcoholic Fatty Liver Disease; Body Weight; Feeding Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study design is an open labelled, randomized, controlled clinical trial, with a ratio 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control group (Active Comparator): All participants in the control group are treated with LED and CBT-based group treatment as described below.
  All participants (control and intervention) receive 2.5-hour sessions of CBT-based group treatment every 4 weeks for 1 year. Participants are randomly assigned to groups of 8-16 participants. Two groups of about the same size start simultaneously.
  The LED phase (from baseline to 24 weeks) consists of 12 weeks with 4 portions/day of liquid meal replacements, for a total of 800-880 kcal/day, followed by a 12-week slow phasing out to a regular diet. Thereafter, an energy-reduced diet (1400-1600 kcal/day) is recommended.
  Interventions: Dietary Supplement: Low energy diet using meal replacements; Behavioral: CBT-based group treatment
- IGB group (Experimental): All participants in the IGB group are treated with LED and CBT-based group treatment as described for the control group.
  Participants in the intervention group are treated with an IGB for 6 months from 6 months from start.
  Interventions: Dietary Supplement: Low energy diet using meal replacements; Behavioral: CBT-based group treatment; Device: Intragastric balloon

INTERVENTIONS:
Dietary Supplement: Low energy diet using meal replacements — The LED phase (from baseline to 24 weeks) consists of 12 weeks with 4 portions/day of liquid meal replacements, for a total of 800-880 kcal/day, followed by a 12-week slow phasing out to a regular diet. Thereafter, an energy-reduced diet (1400-1600 kcal/day) is recommended.
  Other Names: LED
Behavioral: CBT-based group treatment — All participants (control and intervention) receive 2.5-hour sessions of CBT-based group treatment every 4 weeks for 1 year. Participants are randomly assigned to groups of 8-16 participants.
  Other Names: CBT
Device: Intragastric balloon — An IGB (Orbera IGB, Apollo Endosurgery Inc., Austin, Texas, (CE certified)) is set in place endoscopically by a gastroenterologist at Örebro University Hospital, Region Örebro county, and is left in the stomach for 6 months. A proton-pump inhibitor is prescribed to counteract an increased risk to develop a gastric ulcer. During the first 2 weeks, dietary adjustments are necessary to adapt to the IGB. Thereafter, an energy-reduced diet (1400-1600 kcal/day) is recommended identical to the control group. The IGB is removed endoscopically after 6 months IGB treatment.
  Other Names: IGB
  Arms: IGB group

SUMMARY:
In Sweden, approximately 1.3 million adults have obesity. Obesity decreases quality of life (QoL) and increases the risk of diseases such as type 2-diabetes, non-alcoholic fatty liver disease (NAFLD), cancer and cardiovascular diseases. Consequently, weight loss improves QoL and decreases the risk for obesity-related comorbidities.

A treatment combination using a low energy diet (LED) and group treatment based on cognitive behavioral therapy (CBT), leads to 18 percent weight loss after 6 months. Six months treatment with an intragastric balloon (IGB) leads to 13 percent weight loss. However, both treatments are usually followed by weight regain. Combining these treatments has not been studied before but could lead to better weight maintenance.

The hypothesis is that treatment of adults with obesity, with LED, CBT and IGB, leads to greater weight loss after 1 year compared to treatment with LED and CBT only.

The study is a randomized, controlled clinical trial, with a 2-year follow-up. One hundred and ten adults, age 30-65 years, with a BMI of 30-45 kg/m^2 will be included. All participants will receive 6 months of LED, followed by randomization to either 6 months with IGB or a control group without IGB. All participants receive CBT-based group treatment during 12 months and followed up after 2 years.

If the treatment combination of LED, CBT and IGB leads to significant weight loss and improved weight maintenance, increased QoL and reductions of comorbidities and costs of health care are expected. Effects of treatment on eating behavior, NAFLD, physical activity, psychological parameters, the gut microbiota, gut permeability and metabolomics will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 and ≤45 kg/m^2
* Age 30 to 65 years

Exclusion Criteria:

* Participation in an organized weight reduction programme or pharmacological treatment for weight loss within the last 3 months
* Daily use of meal replacement products within the last 3 months
* Previous gastric surgery
* Current gastric, duodenal or oesophageal ulcers
* Inflammatory disease of the gastrointestinal tract including oesophagitis, or specific inflammation such as Crohn's disease
* Known potential upper gastrointestinal bleeding conditions such as gastric or oesophageal varices
* Known structural abnormalities of the pharynx or oesophagus
* Symptoms suggestive for severe gastric motility disorder
* Known hiatus hernia ≥ 5 cm
* Cancer diagnosed within the last 5 years or ongoing treatment for cancer (except non-metastasising skin cancer)
* Known severe heart failure (NYHA 3-4)
* Known chronic obstructive pulmonary disease (FEV1 ≤ 50 percent)
* Kidney failure (eGFR ≤ 30 ml/min)
* Liver failure (liver enzymes more than 3 times the normal threshold)
* Known proliferative retinopathy
* Known or suspected abuse of alcohol or narcotics
* Current or history of systemic treatment with corticosteroids within the last 3 months
* Known myocardial infarction or stroke within the last 6 months
* Current or history of pancreatitis
* Pregnancy, intention to become pregnant or breastfeeding during the study
* Untreated or insufficient treated hypo- or hyperthyroidism
* Current use of anticoagulants: warfarin, apixaban, dabigatran, edoxaban and rivaroxaban
* Current use of thrombocyte aggregation inhibitors: clopidogrel and acetylsalicylic acid
* Known or previous eating disorder
* Antimicrobial treatment within 3 months prior to study may lead to postponed participation
* Regular consumption of probiotic capsules within 1 month prior to study start may lead to postponed participation
* Participants considered to be unsuitable for the study by the investigator (e.g. serious psychiatric disorders, suspected eating disorders)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Weight loss in percent of total body weight | Change from baseline at 12 months
  Total body weight is measured in light indoor clothing without shoes on a calibrated bio-impedance scale.

SECONDARY OUTCOMES:
Weight loss in percent of total body weight | Change from baseline at 6 months
  Total body weight is measured in light indoor clothing without shoes on a calibrated bio-impedance scale.
Weight loss in percent of total body weight at 2-year follow-up | Change from baseline at 24 months
  Two years after treatment start and thus one year after completion of the intervention, participants will be followed up on total body weight. Weight is measured in light indoor clothing without shoes on a calibrated bio-impedance scale.
The proportion of participants with ≥5 percent reduction of total body weight from baseline | 6, 12 and 24 months
  Total body weight is measured in light indoor clothing without shoes on a calibrated bio-impedance scale.
The proportion of participants with ≥10 percent reduction of total body weight from baseline | 6, 12 and 24 months
  Total body weight is measured in light indoor clothing without shoes on a calibrated bio-impedance scale.
The proportion of participants with ≥15 percent reduction of total body weight from baseline | 6, 12 and 24 months
  Total body weight is measured in light indoor clothing without shoes on a calibrated bio-impedance scale.
Effect of treatment on bioelectrical impedance measurement to assess fat mass | Change from baseline at 6, 12 and 24 months
  Bioelectrical impedance analysis is performed with a Body Composition Analyzer BC-420MA. Fatt mass is estimated and results are presented in kilograms.
Effect of treatment on bioelectrical impedance measurement to assess muscle mass | Change from baseline at 6, 12 and 24 months
  Bioelectrical impedance analysis is performed with a Body Composition Analyzer BC-420MA. Muscle mass is estimated and results are presented in kilograms.
Change in waist circumference | Change from baseline at 6, 12 and 24 months
  Waist circumference is measured in centimeters according to the World Health Organization protocol.
Change in 2-hour oral glucose tolerance test | Change from baseline at 6 and 12 months
  Effect on the 2-hour oral glucose tolerance test (OGTT) is measured by analysing glucose (mmol/L) in a fasting blood sample. Thereafter the participant drinks a standardized amount of glucose. After 120 minutes, a blood sample is analyzed again for glucose (mmol/L) .
Change in Hemoglobin A1c | Change from baseline at 6 and 12 months
  Hemoglobin A1c (HbA1c) in mmol/L is analyzed in a fasting blood sample.
Change in serum lipids | Change from baseline at 6 and 12 months
  Total cholesterol, HDL, LDL and triglycerides are analyzed in a fasting blood sample. Results are presented in mmol/L.
Change in insulin | Change from baseline at 6 and 12 months
  Insulin is analyzed in a fasting blood sample and presented in mIE/L.
Change in Homeostatic Model Assessment of Insulin Resistance | Change from baseline at 6 and 12 months
  Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) is calculated using fasting values of insulin and glucose.
Change in kidney function | Change from baseline at 6 and 12 months
  Kidney function is assessed by analysing blood samples for creatinine (µmol/L). The result is used to calculate the estimated glomerular filtration rate (eGFR) using the Lund-Malmö revised calculation. eGFR is presented as mL/min/1,73m^2.
Change in liver transaminases | Change from baseline at 6 and 12 months
  Liver transaminases are measured by analysing alanine transaminase (ALT) and aspartate transaminase (AST) in a fasting blood sample. Data is presented in µkat/L.
Change in thrombocytes | Change from baseline at 6 and 12 months
  Thrombocytes are analyzed in a fasting blood sample and presented as 10*9/L.
Change in blood pressure | Change from baseline at 6 and 12 months
  Blood pressure is measured using a correct cuff size for the circumference of participant's arm after 5 minutes rest in a sitting position.
Effect of treatment on vibration-controlled transient elastography measurement to assess level of liver steatosis and fibrosis | Change from baseline at 6 and 12 months
  Evaluation of NAFLD at baseline and effect of treatment using vibration-controlled transient elastography to detect liver stiffness (in kPa) and determine the steatosis and fibrosis score (0 to 4 there 0 means no steatosis or fibrosis).
Effect of treatment on RAND-36 (SF-36) to measure QoL | Change from baseline at 6, 12 and 24 months
  RAND-36 (SF-36) questionnaire is validated to measure QoL and comprises 36 items measuring eight domains that reflect a wide spectrum of physical and mental health aspects: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health.
Effect of treatment on the Obesity-related Problems scale, version 3 (OPv3) to measure weight-related psychosocial functioning | Change from baseline at 4, 12, 20, 24, 28, 36, 44, 52 and 104 weeks
  OPv3 is validated to measure obesity-specific quality of life with 26 items. OP measures the negative effects of obesity on psychosocial functioning.
Effects of treatment on the Three-Factor Eating Questionnaire-Revised 18 (TFEQ-R18V2) items to measure eating behavior | Change from baseline at 4, 12, 20, 24, 28, 36, 44, 52 and 104 weeks
  The TFEQ-R18V2 is a validated questionnaire to measure three aspects of eating behavior: uncontrolled eating (9 items), cognitive restraint (3 items), and emotional eating (6 items).
Effects of treatment on hunger and satiety | Change from baseline at 4, 12, 20, 24, 28, 36, 44, 52 and 104 weeks
  Hunger and satiety are assessed by a questionnaire with 9 single items on a 5-point Likert scale.
Effect of treatment on 7-day step count to measure physical activity | Change from baseline at 6, 12 and 24 months
  Step count is measured during 7 consecutive days using an accelerometer. The data is completed with questions on water-based activities and cycling on these days.
Effect of treatment on sitting time and physical activity | Change from baseline at 6, 12 and 24 months
  Self-reported data on physical activity will be measured by a validated questionnaire from the National Board of Health and Welfare, Sweden, concerning sitting time and hours of light and moderate activity.
Effect of treatment on the use of medication for glucose lowering treatment, hypertension and hyperlipidemia | Change from baseline at 6, 12 and 24 months
  Effect of treatment on the use of medication for glucose lowering treatment, hypertension and hyperlipidemia is assessed by asking participants at every study contact, if changes in medication have been made. A patient record survey for prescribed medication is performed at 12 and 24 months.
The effect of treatment on the use of health care and absence from work during treatment | Change from baseline at 6, 12 and 24 months
  Health care utilization and absence from work are measured with self-assessment questionnaires. A patient record survey is performed at 12 and 24 months.
Calculation of cost-effectiveness of treatment using multi-variable analysis | Change from baseline at 6, 12 and 24 months
  Cost-effectiveness is analyzed using data on health care utilization, absence from work, use of medication and QoL questionnaires (RAND-36 and OPv3). Data is combined and analyzed together to calculate and report cost-effectiveness. All used measurements are also described above as separate secondary outcome measures.

OTHER OUTCOMES:
Comparison of the calculated risk for liver fibrosis using the fibrosis-4 (FIB-4) calculation to prevalence of liver fibrosis in the study population detected by vibration-controlled transient elastography | At baseline, 6 and 12
  The risk for liver fibrosis is calculated using the FIB-4 calculation (ALT, AST, thrombocytes and age) and compared with results of vibration-controlled transient elastography on prevalence of liver steatosis and fibrosis.
Effect of treatment on lipidomics | Change from baseline at 6 and 12 months
  Evaluation of NAFLD by analysing lipidomic signatures using mass spectrometry based lipidomics.
Change in gut microbiota compositions during treatment with LED, re-introduction of the recommended diet and treatment with IGB | Change from baseline at 2, 4, 6, 9 and 12 months
  Stool samples are taken and will be analyzed for quantitative and qualitative microbial composition by using next generation metagenomic sequencing.
Food frequency questionnaires to evaluate change in dietary intake | Change from baseline, 6 and 12 months
  Food frequency questionnaires (FFQ) will be used to assess dietary intake. This is a common way to evaluate eating habits and, in this way, evaluation of the gut microbiota composition in relation to dietary patterns is possible to assess.
The Bristol Stool Form Scale is used to asses stool form | Change from baseline at 2, 4, 6, 9 and 12 months
  The Bristol Stool Form Scale (BSFS) is used to asses stool form at the same time points as the collection of stool samples. The scale shows 7 pictures of different forms of stool, from watery diarrhea to compact. Participants are asked to choose the most frequent form of stool they have had the past week.
Change in Glucagon-like peptide-1 | Change from baseline at 6 and 12 months
  Glucagon-like peptide-1 (GLP-1) is analysed in a fasting blood sample. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of hormonal parameters in the coming years.
Change in Glucagon-like peptide-2 | Change from baseline at 6 and 12 months
  Glucagon-like peptide-2 (GLP-2) is analysed in a fasting blood sample. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of hormonal parameters in the coming years.
Change in peptide YY | Change from baseline at 6 and 12 months
  Peptide YY (PYY) is analysed in a fasting blood sample. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of hormonal parameters in the coming years.
Change in leptin | Change from baseline at 6 and 12 months
  Leptin is analysed in a fasting blood sample. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of hormonal parameters in the coming years.
Change in ghrelin | Change from baseline at 6 and 12 months
  Ghrelin is analysed in a fasting blood sample. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of hormonal parameters in the coming years.
Change in pro-insulin | Change from baseline at 6 and 12 months
  Pro-insulin is analysed in a fasting blood sample. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of hormonal parameters in the coming years.
Change in C-peptide | Change from baseline at 6 and 12 months
  C-peptide is analysed in a fasting blood sample. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of hormonal parameters in the coming years.
Change in glucagon | Change from baseline at 6 and 12 months
  Glucagon is analysed in a fasting blood sample. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of hormonal parameters in the coming years.
Change in adiponectin | Change from baseline at 6 and 12 months
  Adiponectin is analysed in a fasting blood sample. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of hormonal parameters in the coming years.
Change in glycerol | Change from baseline at 6 and 12 months
  Glycerol is analysed in a fasting blood sample. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of hormonal parameters in the coming years.
Change in free fatty acid | Change from baseline at 6 and 12 months
  Free fatty acid (FFA) is analysed in a fasting blood sample.
Effect of treatment on highly sensitive C-reactive protein | Change from baseline at 6 and 12 months
  Highly sensitive C-reactive protein (hs-CRP) is analysed in mg/L as a measure for inflammation.
  Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of inflammatory parameters in the coming years.
Effect of treatment on Interleukin-6 | Change from baseline at 6 and 12 months
  Interleukin-6 (IL-6) is analysed as a measure for inflammation. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of inflammatory parameters in the coming years.
Effect of treatment on Tumor Necrosis Factor-alfa | Change from baseline at 6 and 12 months
  Tumor Necrosis Factor-alfa (TNF-alfa) is analysed as a measure for inflammation. tumor necrosis factor (TNF)-alfa, and Plasminogen activator inhibitor-1 (PAI-1).
  Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of inflammatory parameters in the coming years.
Effect of treatment on Plasminogen Activator Inhibitor-1 | Change from baseline at 6 and 12 months
  Plasminogen activator inhibitor-1 (PAI-1) is analysed as a measure for inflammation.
  Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of inflammatory parameters in the coming years.
Effect of treatment on metabolomics | Change from baseline at 6 and 12 months
  Changes in metabolomics are assessed by mass spectrometry based approaches for global analysis of molecular lipids (lipidomics) and polar metabolites. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of metabolic parameters in the coming years.
Effect of treatment on Zonulin | Change from baseline at 6 and 12 months
  Zonulin is analysed in a fasting blood sample as a measure for gut permeability. Extra plasma and serum will be collected in a biobank to be able to make use of expected new developed and validated analysis of gut permeability in the coming years.
Gastrointestinal Symptom Rating Scale to assess gastrointestinal symptoms | Baseline, 4, 12, 20, 24, 28, 36, 44 and 52 weeks
  The Gastrointestinal Symptom Rating Scale (GSRS) is an instrument with 15-items validated to assess gastro-intestinal (GI) symptoms associated with GI disorders. It contains 5 subscales (Reflux, Diarrhea, Constipation, Abdominal Pain, and Indigestion Syndrome). The scores per subscale range from 1 to 7. Higher scores represent more discomfort.
Visceral Sensitivity Index to assess fear of gastrointestinal symptoms | Baseline, 4, 12, 20, 24, 28, 36, 44 and 52 weeks
  The Visceral Sensitivity Index (VSI) measures GI symptom-specific anxiety and comprises 15 items.
Nepean Dyspepsia Index to assess dyspepsia | Baseline, 4, 12, 20, 24, 28, 36, 44 and 52 weeks
  The Short form-Nepean dyspepsia index measures upper GI symptoms with 10 items.
Rome IV criteria to assess symptoms for irritable bowel syndrome | Baseline, 6 and 12 months
  Rome IV is a diagnostic questionnaire for functional GI disorders, and comprises of 89 items in a flowchart.
13C Spirulina Breath test to assess gastric emptying rate in participants randomized to IGB treatment | 1 to 28 days before IGB placement
  Gastric emptying rate is measured prior to IGB placement in participants randomized to IGB. Gastric emptying rate will be measured using the FDA-approved non-invasive, non-radioactive 13C Spirulina Breath test (Cairn Diagnostics, Brentwood, Tennessee, USA).
Analysis of number and causes of early extractions of the gastric balloon to asses tolerability of IGB treatment | 24, 28, 36, 44 and 52 weeks
  The number of participants in need of an early extraction of the IGB, thus prior to 6 months treatment, is assessed. The cause for early removal is assessed.
  Specifically, possible causes for intolerability are assessed by combining data on gastric-emptying, the need for early extraction of the IGB (within 6 months), gastro-intestinal symptoms using 4 questionnaires (GSRS, Rome-IV, VSI and Nepean) and two QoL questionnaires (RAND-36 and OP). All these parameters are also described as separate outcome measures.
Change in Depression Module (PHQ-9) questionnaire | Change from baseline at 4, 12, 20, 24, 28, 36, 44 and 52 weeks
  PHQ-9 is used to assess effect of psychological parameters on treatment results and tolerability. To analyze effect of psychological parameters on treatment results, data analyses will combine this data with treatment effect on weight, gastrointestinal symptoms and QoL.
Change in Anxiety module (GAD-7) questionnaire | Change from baseline at 4, 12, 20, 24, 28, 36, 44 and 52 weeks
  GAD-7 is used to assess effect of psychological parameters on treatment results and tolerability. To analyze effect of psychological parameters on treatment results, data analyses will combine this data with treatment effect on weight, gastrointestinal symptoms and QoL.
Change in Somatic symptom severity ('somatization') module (PHQ-15) questionnaire | Change from baseline at 6 and 12 months
  PHQ-15 is used to assess effect of psychological parameters on treatment results and tolerability.To analyze effect of psychological parameters on treatment results, data analyses will combine this data with treatment effect on weight, gastrointestinal symptoms and QoL.
Pittsburgh Sleep Quality Index to assess sleep quality | Change from baseline at 4, 12, 20, 24, 28, 36, 44 and 52 weeks
  Change in sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI).
Acceptance and Action Questionnaire for Weight-Related Difficulties | Change from baseline at 4, 12, 20, 24, 28, 36, 44 and 52 weeks
  Acceptance and Action Questionnaire for Weight-Related Difficulties (AAQ-W) measures experimental and psychological inflexibility in relation to weight-related feelings, thoughts and actions.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Jendle, Professor, Principal Investigator — johan.jendle@oru.se
Locations (1):
- Medicinmottagning 5/Överviktsenheten, University Hospital Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No